CLINICAL TRIAL: NCT07306663
Title: Sintilimab Combined With Chemotherapy Induction Therapy Followed by Concurrent Chemoradiotherapy vs. Concurrent Chemoradiotherapy for Esophageal Cancer: A Randomized Controlled Phase Ⅲ Clinical Study
Brief Title: Sintilimab Combined With Chemotherapy Induction Therapy Followed by CCRT vs. CCRT for Esophageal Cancer: A Randomized Controlled Phase Ⅲ Clinical Study
Acronym: ESO-Nanjing7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Collaborators: Beijing Bethune Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Ye jinjun, Chief Physician, Department of Radiation Oncology, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Nanjing7
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sintilimab; Carboplatin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction group (Experimental): Patients receive induction therapy with sintilimab plus 3-weekly paclitaxel/carboplatin for 2 cycles, followed by concurrent chemoradiotherapy (weekly paclitaxel/carboplatin plus radiotherapy).
  Interventions: Biological: Sintilimab; Drug: 3-Weekly Paclitaxel plus Carboplatin (TC) Chemotherapy; Drug: Weekly TC Chemotherapy; Radiation: Definitive Radiotherapy
- Standard group (Active Comparator): Patients receive concurrent chemoradiotherapy (weekly paclitaxel/carboplatin with radiotherapy), followed by 2 cycles of consolidation chemotherapy (4-weekly paclitaxel/carboplatin).
  Interventions: Drug: Weekly TC Chemotherapy; Drug: Four-Weekly TC Consolidation Chemotherapy; Radiation: Definitive Radiotherapy

INTERVENTIONS:
Biological: Sintilimab — 200mg, once every three weeks, administered before concurrent chemoradiotherapy.
  Arms: Induction group
Drug: 3-Weekly Paclitaxel plus Carboplatin (TC) Chemotherapy — Three-weekly induction chemotherapy regimen: Paclitaxel (135 mg/m², d1) + Carboplatin (AUC=5, d1), administered every 21 days.
  Arms: Induction group
Drug: Weekly TC Chemotherapy — Paclitaxel (50 mg/m², intravenous infusion on Day 1 of each week) combined with Carboplatin (AUC 2, intravenous infusion on Day 1 of each week), administered for 5 consecutive weeks as part of concurrent chemoradiotherapy.
Drug: Four-Weekly TC Consolidation Chemotherapy — Four-weekly consolidation chemotherapy regimen: Paclitaxel (175 mg/m², intravenous infusion on Day 1) combined with Carboplatin (AUC 5, intravenous infusion on Day 1), administered every 28 days for 2 cycles following concurrent chemoradiotherapy.
  Arms: Standard group
Radiation: Definitive Radiotherapy — Definitive radiotherapy administered at a total dose of 50.4 Gy in 28 daily fractions (1.8 Gy per fraction) over approximately 5.5 weeks, delivered concurrently with weekly chemotherapy.

SUMMARY:
The objective of this clinical trial is to determine whether the addition of immunotherapy combined with chemotherapy before chemoradiotherapy can increase the survival rate of patients with esophageal cancer. It will also assess the safety of this regimen. The primary questions it aims to answer include:

* Can the addition of immunotherapy combined with chemotherapy before chemoradiotherapy reduce the rate of disease recurrence among participants?
* What adverse reactions will participants experience during the treatment process?
* Compared with traditional chemoradiotherapy, will this regimen extend the survival period of participants?

Participants will:

* Undergo two cycles of immunotherapy combined with chemotherapy, administered every three weeks, followed by concurrent chemoradiotherapy, which includes 28 sessions of radiotherapy and five sessions of chemotherapy during the concurrent period; or proceed directly to concurrent chemoradiotherapy, and then receive two cycles of chemotherapy after the completion of radiotherapy, administered once a month.
* Undergo regular tests and examinations to evaluate efficacy and safety.
* Record symptoms that occur during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and provide written informed consent;
2. Age 18-75 years, regardless of gender;
3. Histologically or cytologically confirmed esophageal squamous cell carcinoma;
4. Patients with inoperable esophageal cancer;
5. Clinical stage Ⅱ-ⅣA (AJCC 8th edition esophageal cancer staging system, including stage ⅣB with supraclavicular lymph node metastasis but excluding other distant metastatic stage ⅣB);
6. ECOG performance status 0-1;
7. Expected survival ≥ 3 months;
8. No severe dysfunction of hematopoietic, cardiac, pulmonary, hepatic, or renal systems, nor immune deficiency; Neutrophils ≥ 1.5×10⁹/L; hemoglobin ≥ 9 g/dL; platelets ≥ 100×10⁹/L; total bilirubin ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; creatinine ≤ 1.5 × ULN.

Exclusion Criteria:

1. Esophageal perforation or hematemesis;
2. Active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (patients with hypothyroidism stable on hormone replacement therapy for ≥4 weeks with TSH/FT4 within normal range may be included); additionally, patients who have used immunosuppressants within 28 days will be excluded, except for steroid use for managing chemoradiation-related toxicities;
3. Previous or ongoing treatment with other types of PD-1 antibodies, or prior immunotherapy targeting PD-1/PD-L1;
4. Known allergic reaction to macromolecular protein drugs or sintilimab or any of its formulation components;
5. Uncontrolled cardiac disease or clinical symptoms, such as: a. heart failure of NYHA class II or above; b. unstable angina; c. myocardial infarction within the past year; d. supraventricular or ventricular arrhythmias requiring clinical intervention;
6. Congenital or acquired immunodeficiency (e.g., HIV infection), active hepatitis B (HBV-DNA ≥ 10⁴ copies/mL), hepatitis C (positive HCV antibody with HCV-RNA above the lower limit of detection), or active tuberculosis;
7. Active infection, or unexplained fever (body temperature >38.5℃) within 2 weeks prior to screening (fever judged by the investigator to be due to the tumor itself may be allowed);
8. Male or female participants of childbearing potential who refuse to use contraception during the study; or female patients who are pregnant or breastfeeding;
9. Other conditions judged by the investigator that may lead to premature termination of the study, such as co-existing severe diseases (including psychiatric disorders) requiring combined treatment, or family/social factors that may affect participant safety or integrity of the trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 242 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | From the date of randomization to 3 years or until death, whichever comes first.

SECONDARY OUTCOMES:
Progression-free survival | From the date of randomization to 3 years or until disease progression or death, whichever occurs first.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | For the duration of treatment plus 30 days after the last dose.
Objective response rate | One month after the completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Ye, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided